CLINICAL TRIAL: NCT01645124
Title: A Large-scale Trial Testing the Intensity of CYTOreductive Therapy to Prevent Cardiovascular Events In Patients With Polycythemia Vera (PV)
Brief Title: Large-scale Trial Testing the Intensity of CYTOreductive Therapy in Polycythemia Vera (PV)
Acronym: CYTO-PV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low accrual rate not allowing planned sample size leads to a futility condition
Sponsor: Consorzio Mario Negri Sud (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government); A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FARM6YNXAN
Record Dates: First submitted 2012-07-17; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-05

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia; Hematocrit; Thrombosis
MeSH Terms: conditions — Polycythemia Vera; Polycythemia; Thrombosis | interventions — Hydroxyurea; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cytoreduction for HCT < 45% (Active Comparator): Patients will be treated with phlebotomy and/or HU more intensively, with the goal to reach and maintain the target of hematocrit(HCT)below 45%. Phlebotomy should be performed initially by removing 250-500 ml of every other day or twice a week until the target HCT is obtained. Hydroxyurea (HU)should be administered initially at a dose of 0.5-1.0 g daily. Blood counts at regular intervals (monthly) will establish the frequency of future phlebotomies with the goal to maintain the target HCT. Supplemental iron therapy should not be given. Low-dose aspirin is the standard antithrombotic therapy in PV and will be administered to all patients with no contraindications to aspirin.
  Interventions: Drug: Hydroxyurea; Procedure: Phlebotomy
- Cytoreduction for HCT between 45 and 50% (Experimental): Patients will be treated with phlebotomy and/or HU less intensively, with the goal to reach and maintain the target of hematocrit(HCT)between 45% and 50%. Phlebotomy should be performed initially by removing 250-500 ml of every other day or twice a week until the target HCT is obtained. Hydroxyurea (HU)should be administered initially at a dose of 0.5-1.0 g daily. Blood counts at regular intervals (monthly) will establish the frequency of future phlebotomies with the goal to maintain the target HCT. Supplemental iron therapy should not be given. Low-dose aspirin is the standard antithrombotic therapy in PV and will be administered to all patients with no contraindications to aspirin.
  Interventions: Drug: Hydroxyurea; Procedure: Phlebotomy

INTERVENTIONS:
Drug: Hydroxyurea
Procedure: Phlebotomy

SUMMARY:
CYTO-PV is a phase III Prospective, Randomized, Open-label, with Blinded Endpoint evaluation (PROBE), multi-center, clinical trial in patients with diagnosis of Polycythemia vera (PV) treated at the best of recommended therapies (e.g.adequate control of standard cardiovascular risk factors). Irrespective of randomized interventions, all patients will be administered low-dose aspirin (when not contraindicated), i.e.the standard antithrombotic treatment in PV patients.

The purpose of this study to demonstrate that a more intensive cytoreductive therapy, plus low-dose aspirin when not contraindicated, with phlebotomy and/or hydroxyurea (HU), aimed at maintaining hematocrit (HCT) < 45% is more effective than a less intensive cytoreduction (either with phlebotomy or HU plus low-dose aspirin when not contraindicated) maintaining HCT in the range of 45-50% in the reduction of CV deaths plus thrombotic events (stroke, acute coronary syndrome [ACS], transient ischemic attack [TIA], pulmonary embolism [PE], splanchnic thrombosis, deep vein thrombosis [DVT], and any other clinically relevant thrombotic event), in patients with Polycythemia Vera treated at the best of recommended therapies (e.g. adequate control of standard cardiovascular risk factors).

DETAILED DESCRIPTION:
Polycythemia vera (PV) is a chronic myeloproliferative disorder characterized by clonal proliferation of hematopoietic progenitors resulting in expansion of the erythrocyte mass, and its clinical course is affected by cardiovascular events, the main cause of morbidity and mortality. Arterial thrombotic events are predominant, particularly large vessel arterial events including cerebrovascular accidents, myocardial infarction, and peripheral arterial occlusion. Based on the complex relationship between thrombosis, hematocrit, and parameters of tissue perfusion and blood viscosity, the latter has been proved to be an exponential function of the hematocrit. Red cell aggregation increases at high hematocrit (HCT) levels, creating the potential for vascular stasis. As a result, enhanced interplay between platelet, leukocytes and vessel wall increases the risk of thrombosis.

Considering the lack of effective therapeutic strategy targeted at the mutated allele JAK2V617F, there is no known treatment that eradicates the abnormal clone, apart from anecdotal cases of bone marrow transplantation. Cytoreductive treatment by phlebotomy or chemotherapy, however, has dramatically reduced the number of thrombotic complications and substantially improved survival and today there is agreement that the goal of cytoreductive treatment should be to keep the HCT value below 0.45 in all PV patients.

This was suggested on the basis of a small, retrospective study of PV that more than 30 years ago showed a progressive increase in the incidence of vascular occlusive episodes at HCT levels higher than 44% and in patients treated according to the drugs and the therapeutic tenets of the time. However no clinical trial has confirmed such findings. The results of the two largest prospective studies currently available (namely PVSG-1 and ECLAP) suggest no difference in the risk of thrombosis among patients kept at HCT below 50%.

An association between relevant outcome events (namely. thrombotic events, mortality, and haematological progression) and HCT in the evaluable range of 40-55% was found in the ECLAP population neither in the multivariate analysis at baseline nor in the time-dependent multivariate analysis. The ECLAP trial demonstrated the antithrombotic efficacy of low-dose aspirin in this setting and the use of this therapy in clinical practice is likely to decrease meaningfully, though not eliminate, the high risk of thrombosis of PV patients.

In conclusion, the high incidence of thrombotic events irrespective of low-dose aspirin administration as well as of haematological transformation in the long term which have been shown in PV patients study suggest the need to investigate in depth the benefit/risk profile of current therapeutic options for cytoreductive therapy. CYTO-PV is aimed at assessing the benefit risk profile of cytoreductive therapy with phlebotomy and/or HU aimed at maintaining HCT < 45% Vs. maintaining HCT in the range 45-50%. It is an independent, investigator-generated pragmatic trial with broad selection criteria to mimic clinical practice in order to strengthen the transferability of its results to the population of PV patients; it has been designed to be conducted, without need of special facilities, in the framework of the Italian Group of hematologic Adult diseases ("GIMEMA"). The optimization of therapeutic management of PV patients will allow to improve the prognosis of PV patients, the allocation of the resources the Italian National Health Service (IHS), and the knowledge about the benefit/risk profile of pharmacological cytoreduction in PV

ELIGIBILITY:
Inclusion Criteria:

Males and females aged 18 years or more are eligible for the study if they meet all the following inclusion criteria:

* New diagnosis of PV according to WHO 2007 diagnostic criteria including Jak 2 V617F mutation status;
* Old diagnosis of PV confirmed with JAK-2 positivity and clinical course of the disease;
* Ability and willingness to comply with all study requirements;
* Written informed consent (obtained before any study specific procedure).

Exclusion Criteria:

* Pregnant or lactating women or women of childbearing potential who are not protected from pregnancy by an accepted method of contraception;
* Known hypersensitivity or contraindication to study treatments;
* Significant liver (AST or ALT > 2.5 times ULN) or renal disease (creatinine > 2 mg/ml);
* Presence of any life-threatening condition or of any disease (e.g. cancer) that is likely to significantly shorten life expectancy;
* History of active substance or alcohol abuse within the last year;
* Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety or be associated with poor adherence to the protocol - Baseline and FUP visits schedule and assessments
* Logistic problem related to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2008-05; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Reduction of PEP (Primary End Point)defined as CV deaths plus thrombotic events | Expected average of 5 years
  To demonstrate that in patients with PV treatment with aggressive cytoreductive therapy aimed at maintaining HCT < 45% is more effective than cytoreductive therapy aimed at maintaining HCT between 45 and 50% in the reduction CV deaths plus thrombotic events (PEP: stroke, acute coronary syndrome [ACS], transient ischemic attack [TIA], pulmonary embolism [PE], abdominal thrombosis, deep vein thrombosis [DVT], and peripheral arterial thrombosis). The minimum clinically relevant beneficial effect is set at a 30% reduction of risk of the PEP.

SECONDARY OUTCOMES:
PEP plus minor thrombosis, hospitalization and malignancy | Expected average of 5 years
  The events included in the PEP, arterial and venous thrombosis, major and minor thrombosis as well as hospitalization for any reason, hospitalization for CV reason, malignancy and PV-related malignancy (progression to myelofibrosis, myelodysplastic or leukemic transformation) will be analyzed separately to assess the full benefit/risk profile of experimental treatments.

OTHER OUTCOMES:
Aadverse Events | Expected average of 5 years
  Background knowledge suggests that no specific safety precautions are to be adopted for phlebotomy and HU administration. However, both pragmatic reasons and the consideration of the clinical condition under study (see: age, comorbidity, polytherapy) support the decision to adopt a generalized policy of surveillance specifically on:
  * Hypotension or syncope after phlebotomy;
  * renal dysfunction (creatinine);
  * liver dysfunction (ALT, AST, symptoms);
  * White blood cell count;
  * Platelet count;
  * Bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Tiziano Barbui, MD, Study Chair — A.O. Ospedale Papa Giovanni XXIII
Locations (26):
- Italy (26):
  - Azienda Ospedaliera Universitaria Ospedali Riuniti di Ancona, Ancona, Ancona
  - Azienda Ospedaliera Universitaria Ospedale Consorziale Policlinico di Bari, Bari, Bari
  - Azienda Ospedali Riuniti di Bergamo, Bergamo, Bergamo
  - Azienda Unità Sanitaria Locale di Brindisi BR/1- Ospedale "Di Summa - Perrino", Brindisi, Brindisi
  - Ospedale Armando Businco, Cagliari, Cagliari
  - Azienda Ospedaliera Universitaria-'Policlinico- Vittorio Emanuele'-Ospedale Ferrarotto Alessi di Catania, Catania, Catania
  - Azienda Ospedaliera S. Croce e Carle di Cuneo, Cuneo, Cuneo
  - Azienda Ospedaliera Universitaria Careggi di Firenze, Florence, Firenze
  - IRCCS Ospedale Casa Sollievo della Sofferenza di San Giovanni Rotondo, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Universitaria Policlinico Martino di Messina, Messina, Messina
  - Fondazione IRCSS Cà Granda- Ospedale Maggiore Policlinico, Milan, Milano
  - Ospedale S.Raffaele, Milan, Milano
  - Ospedale S.Gerardo di Monza, Monza, Monza
  - Azienda Ospedaliera Universitaria'Maggiore della Carità' di Novara, Novara, Novara
  - Università di Padova, Padua, Padova
  - Azienda Ospedaliero-Universitaria Policlinico Giaccone di Palermo, Palermo, Palermo
  - IRCCS Policlinico S. Matteo di Pavia, Pavia, Pavia
  - Azienda Ospedaliera S. Salvatore, Presidio San Salvatore Muraglia, Pesaro, Pesaro
  - IRCCS Centro di Riferimento Oncologico di Basilicata (CROB), Rionero in Vulture, Potenza
  - AUSL 4 Prato, Ospedale "Misericordia e Dolce" di Prato, Prato, Prato
  - Ospedale di S.Maria Nuova, Reggio Emilia, Reggio Emilia
  - IRCCS Istituto Regina Elena (IFO), Roma, Roma
  - Università degli Studi di Roma "La Sapienza", Roma, Roma
  - Policlinico Universitario Gemelli di Roma, Roma, Roma
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga di Orbassano, Orbassano, Torino
  - Ospedale San Bortolo di Vicenza, Vicenza, Vicenza

REFERENCES:
- [Derived] Marchioli R, Finazzi G, Specchia G, Cacciola R, Cavazzina R, Cilloni D, De Stefano V, Elli E, Iurlo A, Latagliata R, Lunghi F, Lunghi M, Marfisi RM, Musto P, Masciulli A, Musolino C, Cascavilla N, Quarta G, Randi ML, Rapezzi D, Ruggeri M, Rumi E, Scortechini AR, Santini S, Scarano M, Siragusa S, Spadea A, Tieghi A, Angelucci E, Visani G, Vannucchi AM, Barbui T; CYTO-PV Collaborative Group. Cardiovascular events and intensity of treatment in polycythemia vera. N Engl J Med. 2013 Jan 3;368(1):22-33. doi: 10.1056/NEJMoa1208500. Epub 2012 Dec 8. PMID 23216616